CLINICAL TRIAL: NCT00829010
Title: Primary and Booster Vaccination Course in Human Immunodeficiency Virus (HIV) Infected Infants, HIV Exposed Uninfected Infants and Unexposed Uninfected Infants Receiving the Pneumococcal Vaccine GSK 1024850A.
Brief Title: Primary and Booster Vaccination Study With a Pneumococcal Vaccine in HIV Infected, HIV Exposed Uninfected and HIV Uninfected Children 6 to 10 Weeks of Age.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111634
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Results first posted 2012-07-06 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2017-10

CONDITIONS: Infections, Streptococcal
Keywords: Human Immunodeficiency Virus; Booster vaccination; Safety; Primary vaccination; Pneumococcal vaccine; Immunogenicity; Pneumococcal disease
MeSH Terms: conditions — Streptococcal Infections; Acquired Immunodeficiency Syndrome; Pneumococcal Infections | interventions — RIX4414 vaccine; ZC3H7B protein, human; Poliovirus Vaccine, Oral

ARMS (5):
- HIV+/+ Group (Experimental): Infants born from a HIV positive mother and confirmed as HIV infected. Subjects received 3 primary doses (at 6, 10 & 14 weeks of age, at study Months 0, 1 and 2) and 1 booster dose of Synflorix™ vaccine (at 9 months of age, at study Month 8). Subjects in the group also received 3 primary vaccine doses (at 6, 10 & 14 weeks of age, at study Months 0, 1 and 2) and 1 booster vaccine dose (at 15-18 months of age, at study Month 14) of Tritanrix™-HepB/Hib, 2 vaccine doses of Rotarix™ (at 10 & 14 weeks of age, at study Months 1 and 2), and 2 doses of measles vaccine (9-10 months of age & 15-18 months of age, at study Months 8 and 14). Measles vaccine was not considered as a study vaccine. The Synflorix™ vaccine was administered intramuscularly in the right thigh, the Tritanrix™-HepB/Hib vaccine was administered IM in the left anterolateral thigh during the primary vaccination and in the left anterolateral thigh or left deltoid region during booster vaccination. Rotarix™ was given orally.
  Interventions: Biological: Pneumococcal vaccine GSK1024850A; Biological: Tritanrix-HepB/Hib; Biological: measles; Biological: Rotarix; Biological: Local OPV
- HIV+/- Group (Experimental): Infants born from a HIV positive mother and confirmed as HIV exposed uninfected. Subjects received 3 primary doses (at 6, 10 & 14 weeks of age, at study Months 0, 1 and 2) and 1 booster dose of Synflorix™ vaccine (at 9 months of age, at study Month 8). Subjects in the group also received 3 primary vaccine doses (at 6, 10 & 14 weeks of age, at study Months 0, 1 and 2) and 1 booster vaccine dose (at 15-18 months of age, at study Month 14) of Tritanrix™-HepB/Hib, 2 vaccine doses of Rotarix™ (at 10 & 14 weeks of age, at study Months 1 and 2), and 2 doses of measles vaccine (9-10 months of age & 15-18 months of age, at study Months 8 and 14). Measles vaccine was not considered as a study vaccine. The Synflorix™ vaccine was administered IM in the right thigh, the Tritanrix™-HepB/Hib vaccine was administered IM in the left anterolateral thigh during the primary vaccination and in the left anterolateral thigh or left deltoid region during booster vaccination. Rotarix™ was given orally.
  Interventions: Biological: Pneumococcal vaccine GSK1024850A; Biological: Tritanrix-HepB/Hib; Biological: measles; Biological: Rotarix; Biological: Local OPV
- HIV- (3+1) Group (Experimental): Infants born from a HIV negative mother and confirmed as HIV unexposed uninfected. Subjects received 3 primary doses (at 6, 10 & 14 weeks of age, at study Months 0, 1 and 2) and 1 booster dose of Synflorix™ vaccine (at 9 months of age, at study Month 8). Subjects in the group also received 3 primary vaccine doses (at 6, 10 & 14 weeks of age, at study Months 0, 1 and 2) and 1 booster vaccine dose (at 15-18 months of age, at study Month 14) of Tritanrix™-HepB/Hib, 2 vaccine doses of Rotarix™ (at 10 & 14 weeks of age, at study Months 1 and 2), and 2 doses of measles vaccine (9-10 months of age & 15-18 months of age, at study Months 8 and 14). Measles vaccine was not considered as a study vaccine. The Synflorix™ vaccine was administered IM in the right thigh, the Tritanrix™-HepB/Hib vaccine was administered IM in the left anterolateral thigh during the primary vaccination and in the left anterolateral thigh or left deltoid region during booster vaccination. Rotarix™ was given orally.
  Interventions: Biological: Pneumococcal vaccine GSK1024850A; Biological: Tritanrix-HepB/Hib; Biological: measles; Biological: Rotarix; Biological: Local OPV
- HIV- (EPI) Group (Experimental): Infants born from a HIV negative mother and confirmed as HIV unexposed uninfected.Subjects received 3 primary doses of Synflorix™ vaccine (at 6, 10 & 14 weeks of age, at study Months 0, 1 and 2). Subjects in the group also received 3 primary vaccine doses (at 6, 10 & 14 weeks of age, at study Months 0, 1 and 2) and 1 booster vaccine dose (at 15-18 months of age, at study Month 14) of Tritanrix™-HepB/Hib, 2 vaccine doses of Rotarix™ (at 10 & 14 weeks of age, at study Months 1 and 2), and 2 doses of measles vaccine (9-10 months of age & 15-18 months of age, at study Months 8 and 14). Measles vaccine was not considered as a study vaccine. The Synflorix™ vaccine was administered IM in the right thigh, the Tritanrix™-HepB/Hib vaccine was administered IM in the left anterolateral thigh during the primary vaccination and in the left anterolateral thigh or left deltoid region during booster vaccination. Rotarix™ was given orally.
  Interventions: Biological: Pneumococcal vaccine GSK1024850A; Biological: Tritanrix-HepB/Hib; Biological: measles; Biological: Rotarix; Biological: Local OPV
- HIV- (2+1) Group (Experimental): Infants born from a HIV negative mother and confirmed as HIV unexposed uninfected.Subjects received 2 primary doses (at 6 & 14 weeks of age at study Months 0 and 2) and 1 booster dose of Synflorix™ vaccine (at 9 months of age, at study Month 8). Subjects in the group also received 3 primary vaccine doses (at 6, 10 & 14 weeks of age, at study Months 0, 1 and 2) and 1 booster vaccine dose (at 15-18 months of age, at study Month 14) of Tritanrix™-HepB/Hib, 2 vaccine doses of Rotarix™ (at 10 & 14 weeks of age, at study Months 1 and 2), and 2 doses of measles vaccine (9-10 months of age & 15-18 months of age, at study Months 8 and 14). Measles vaccine was not considered as a study vaccine. The Synflorix™ vaccine was administered IM in the right thigh, the Tritanrix™-HepB/Hib vaccine was administered IM in the left anterolateral thigh during the primary vaccination and in the left anterolateral thigh or left deltoid region during booster vaccination. Rotarix™ was given orally.
  Interventions: Biological: Pneumococcal vaccine GSK1024850A; Biological: Tritanrix-HepB/Hib; Biological: measles; Biological: Rotarix; Biological: Local OPV

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK1024850A — Intramuscular injection, administered as 3 or 4 doses
Biological: Tritanrix-HepB/Hib — Intramuscular injection, 4 doses
  Other Names: DTPw-HBV/Hib
Biological: measles — Intramuscular injection, 2 doses
Biological: Rotarix — Oral, 2 doses
  Other Names: HRV; Human rotavirus
Biological: Local OPV — Oral 4 doses. Given at any time during the study, routinely given concurrently with DTPw-HBV/Hib vaccine
  Other Names: oral poliovirus vaccine

SUMMARY:
The purposes of this study:

* To evaluate the immunogenicity, safety and reactogenicity of pneumococcal vaccine GSK1024850A in HIV infected infants, HIV exposed uninfected infants and HIV unexposed uninfected infants following a 3-dose primary vaccination at 6, 10 and 14 weeks of age and following booster vaccination at 9-10 months of age.
* To evaluate the immunogenicity, safety and reactogenicity of pneumococcal vaccine GSK1024850A in HIV unexposed uninfected infants receiving either a 3-dose primary vaccination according to the EPI vaccination schedule at 6, 10 and 14 weeks of age with or without booster vaccination at 9-10 months of age or a 2-dose primary vaccination at 6 and 14 weeks of age followed by booster vaccination at 9-10 months of age.
* This study also aims to assess the impact of the pneumococcal vaccine GSK1024850A on nasopharyngeal carriage of S. pneumoniae and H. influenzae up to 24 months of age in all study participants.

DETAILED DESCRIPTION:
This protocol posting has been updated according to Protocol amendment 1, December 08

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between, and including 6-10 weeks of age at the time of the first vaccination.
* Subjects for whom the investigator believes that their parent(s)/guardian(s) can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/guardian(s) of the child/ward.
* Free of any known or suspected health problems (as established by medical history and clinical examination before entering into the study).

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of the study vaccines, or planned use during the study period.
* A family history of hereditary immunodeficiency other than HIV infection.
* Major congenital defects or serious chronic illness other than HIV infection.
* For HIV infected infants: Moderately and severely symptomatic: stages III and IV according to latest version of WHO classification.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Previous vaccination against diphtheria, tetanus, pertussis, hepatitis B, Haemophilus influenzae type b, and/or Streptococcus pneumoniae.
* History of, or intercurrent, diphtheria, tetanus, pertussis, and Haemophilus influenzae type b disease.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of any neurological disorders or seizures.
* Acute disease at the time of enrolment.
* Babies for which weight for age is < 3rd percentile at Visit 1, using standard growth charts, with the exception of HIV infected infants for which the decision of enrolment was left to the investigator's discretion.
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the gastrointestinal (GI) tract, intussusception (IS) or other medical condition determined to be serious by the investigator.
* Gastroenteritis within 7 days preceding the study vaccine administration (warrants deferral of vaccination).

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 489 (Actual)
Dates: Start 2009-02-17; Primary Completion 2011-06-13 (Actual); Study Completion 2012-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Soweto, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Izu A, Koen A, Jose L, Cutland C, de Gouveia L, von Gottberg A, Groome MJ, Jones S, Madhi SA. Persistence of Antibodies at Three, Four and Five Years of Age to Ten-valent Pneumococcal Polysaccharide Protein D-conjugate Vaccine in South African Children According to HIV Status. Pediatr Infect Dis J. 2026 Feb 1;45(2):173-180. doi: 10.1097/INF.0000000000005050. Epub 2025 Dec 3. PMID 41495936
- [Derived] Nunes MC, Moreira M, Koen A, van Niekerk N, Jose L, Cutland CL, Francois N, Schoonbroodt S, Ruiz-Guinazu J, Yarzabal JP, Borys D, Schuerman L, Madhi SA. Bacterial nasopharyngeal carriage following infant immunization with pneumococcal conjugate vaccines according to a 2+1 schedule in children in South Africa: an exploratory analysis of two clinical trials. Expert Rev Vaccines. 2020 Dec;19(12):1177-1189. doi: 10.1080/14760584.2020.1853533. Epub 2020 Dec 21. PMID 33245004
- [Derived] Madhi SA, Moreira M, Koen A, van Niekerk N, de Gouveia L, Jose L, Cutland CL, Francois N, Schoonbroodt S, Ruiz-Guinazu J, Yarzabal JP, Borys D, Schuerman L. Impact of HIV status and vaccination schedule on bacterial nasopharyngeal carriage following infant immunisation with the pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine in South Africa. Vaccine. 2020 Feb 28;38(10):2350-2360. doi: 10.1016/j.vaccine.2020.01.062. Epub 2020 Feb 5. PMID 32035706
- [Derived] Madhi SA, Koen A, Jose L, Moreira M, van Niekerk N, Cutland C, Francois N, Ruiz-Guinazu J, Yarzabal JP, Borys D, Schuerman L. Immunization with 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) according to different schedules in infants in South Africa: a phase III trial. Expert Rev Vaccines. 2017 Jun;16(6):641-656. doi: 10.1080/14760584.2017.1321990. PMID 28425818
- [Derived] Madhi SA, Koen A, Jose L, van Niekerk N, Adrian PV, Cutland C, Francois N, Ruiz-Guinazu J, Yarzabal JP, Moreira M, Borys D, Schuerman L. Vaccination with 10-valent pneumococcal conjugate vaccine in infants according to HIV status. Medicine (Baltimore). 2017 Jan;96(2):e5881. doi: 10.1097/MD.0000000000005881. PMID 28079828
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 111634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111634 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The oral poliovirus vaccine could be given at any time during the study (routinely given concurrently with Tritanrix™-HepB/Hib vaccine) but was not considered as study vaccine. Out of the 489 subjects enrolled in the study, 484 subjects were assigned to a study group and received vaccination.
Pre-assignment Details: The study included 3 populations defined based on the human immunodeficiency virus status of the mother and the infant. Infant born from:
  * a HIV positive mother and HIV infected at Month 0 = HIV+/+.
  * a HIV positive mother and HIV exposed uninfected at screening = HIV+/-.
  * a HIV negative mother and HIV unexposed uninfected at Month 0 = HIV-
Groups:
- HIV+/+ Group: Infants born from a HIV positive mother and confirmed as HIV infected. Subjects received 3 primary doses (at 6, 10 & 14 weeks of age, at study Months 0, 1 and 2) and 1 booster dose of Synflorix™ vaccine (at 9 months of age, at study Month 8). Subjects in the group also received 3 primary vaccine doses (at 6, 10 & 14 weeks of age, at study Months 0, 1 and 2) and 1 booster vaccine dose (at 15-18 months of age, at study Month 14) of Tritanrix™-HepB/Hib, 2 vaccine doses of Rotarix™ (at 10 & 14 weeks of age, at study Months 1 and 2), and 2 doses of measles vaccine (9-10 months of age & 15-18 months of age, at study Months 8 and 14). Measles vaccine was not considered as study vaccine. The Synflorix™ vaccine was administered intramuscularly (IM) in the right thigh, the Tritanrix™-HepB/Hib vaccine was administered IM in the left anterolateral thigh during the primary vaccination and in the left anterolateral thigh or left deltoid region during booster vaccination. Rotarix™ was given orally.
- HIV- (3+0) Group: Infants born from a HIV negative mother and confirmed as HIV unexposed uninfected.Subjects received 3 primary doses of Synflorix™ vaccine (at 6, 10 & 14 weeks of age, at study Months 0, 1 and 2). Subjects in the group also received 3 primary vaccine doses (at 6, 10 & 14 weeks of age, at study Months 0, 1 and 2) and 1 booster vaccine dose (at 15-18 months of age, at study Month 14) of Tritanrix™-HepB/Hib, 2 vaccine doses of Rotarix™ (at 10 & 14 weeks of age, at study Months 1 and 2), and 2 doses of measles vaccine (9-10 months of age & 15-18 months of age, at study Months 8 and 14). Measles vaccine was not considered as a study vaccine. The Synflorix™ vaccine was administered IM in the right thigh, the Tritanrix™-HepB/Hib vaccine was administered IM in the left anterolateral thigh during the primary vaccination and in the left anterolateral thigh or left deltoid region during booster vaccination. Rotarix™ was given orally.
Period: Overall Study
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Started | 83 | 101 | 100 | 100 | 100
Completed | 73 | 92 | 97 | 92 | 98
Not Completed | 10 | 9 | 3 | 8 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0 | 0
Not completed — Fatality | 5 | 4 | 0 | 3 | 0
Not completed — Migrated/Moved from study area | 3 | 4 | 0 | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group | Total
Number analyzed (Participants) | 83 | 101 | 100 | 100 | 100 | 484
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 6.6 (0.92) | 6.3 (0.65) | 6.1 (0.41) | 6.1 (0.35) | 6.1 (0.29) | 6.2 (0.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 47 | 58 | 50 | 47 | 251
  Male | 34 | 54 | 42 | 50 | 53 | 233

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-pneumococcal Vaccine Serotype Antibody Concentrations Equal to or Above 0.20 Microgram Per Millilitre (µg/mL).
Description: Pneumococcal vaccine serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
Time Frame: 1 month following primary immunization (post-Dose 3 at Month 3 for the HIV+/+ Group, HIV+/- Group, HIV- (3+1) Group, HIV- (3+0) Group and post-Dose 2 at Month 3 for the HIV- (2+1) Group)
Population: The According-To-Protocol cohort for immunogenicity included evaluable subjects for whom data concerning immunogenicity outcome measures were available. This included subjects for whom assay results were available for antibodies against at least 1 study vaccine antigen component post dose II or III, as applicable, or after booster vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 70 | 91 | 93 | 94 | 97
Participants
  Anti-1 | 69 | 90 | 93 | 94 | 96
  Anti-4: number analyzed (Participants) | 70 | 91 | 93 | 93 | 97
  Anti-4 | 69 | 90 | 93 | 93 | 96
  Anti-5 | 70 | 90 | 93 | 94 | 95
  Anti-6B: number analyzed (Participants) | 70 | 91 | 93 | 93 | 97
  Anti-6B | 61 | 80 | 74 | 83 | 80
  Anti-7F | 69 | 90 | 93 | 94 | 96
  Anti-9V | 68 | 90 | 93 | 94 | 92
  Anti-14: number analyzed (Participants) | 70 | 91 | 93 | 93 | 97
  Anti-14 | 69 | 90 | 93 | 93 | 95
  Anti-18C: number analyzed (Participants) | 69 | 91 | 93 | 94 | 97
  Anti-18C | 69 | 90 | 93 | 94 | 95
  Anti-19F: number analyzed (Participants) | 70 | 91 | 93 | 93 | 96
  Anti-19F | 68 | 90 | 93 | 93 | 94
  Anti-23F: number analyzed (Participants) | 70 | 91 | 93 | 93 | 97
  Anti-23F | 63 | 84 | 83 | 84 | 84

2. Secondary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes.
Description: Concentrations were given in microgram per millilitre (µg/mL) and were expressed in geometric mean antibody concentrations. Pneumococcal vaccine serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Data were collected post-Dose 3 at Month 3 and post-Dose 4 at Month 9 for the HIV+/+, HIV+/- and HIV- (3+1) groups, post-Dose 3 at Month 3 and at Month 9 for HIV- (3+0) group, and post-Dose 2 at Month 3 and post-Dose 3 at Month 9 for the HIV- (2+1) Group. The cut-off of the assay is 0.05 µg/mL.
Time Frame: At Month 3 and Month 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/ml
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 70 | 91 | 93 | 94 | 97
µg/ml
  Anti-1 [Month 3] | 4.00 [3.30 to 4.84] | 3.85 [3.26 to 4.55] | 3.36 [2.91 to 3.88] | 4.65 [3.91 to 5.53] | 3.33 [2.85 to 3.88]
  Anti-1 [Month 9]: number analyzed (Participants) | 66 | 89 | 93 | 93 | 97
  Anti-1 [Month 9] | 6.64 [5.22 to 8.46] | 8.64 [7.09 to 10.53] | 5.38 [4.47 to 6.48] | 0.72 [0.58 to 0.88] | 5.14 [4.42 to 5.97]
  Anti-4 [Month 3]: number analyzed (Participants) | 70 | 91 | 93 | 93 | 97
  Anti-4 [Month 3] | 3.67 [2.81 to 4.80] | 3.14 [2.60 to 3.80] | 2.71 [2.28 to 3.21] | 3.77 [3.09 to 4.60] | 2.28 [1.90 to 2.75]
  Anti-4 [Month 9]: number analyzed (Participants) | 66 | 89 | 93 | 93 | 97
  Anti-4 [Month 9] | 6.97 [5.72 to 8.50] | 8.04 [6.69 to 9.68] | 6.07 [5.09 to 7.24] | 1.07 [0.86 to 1.34] | 4.92 [4.16 to 5.81]
  Anti-5 [Month 3] | 4.99 [4.00 to 6.23] | 4.79 [3.96 to 5.79] | 4.41 [3.79 to 5.13] | 5.71 [4.84 to 6.75] | 3.45 [2.85 to 4.16]
  Anti-5 [Month 9]: number analyzed (Participants) | 66 | 89 | 93 | 93 | 97
  Anti-5 [Month 9] | 7.86 [6.25 to 9.89] | 9.48 [7.84 to 11.46] | 8.05 [6.70 to 9.66] | 1.44 [1.16 to 1.77] | 6.96 [5.89 to 8.22]
  Anti-6B [Month 3]: number analyzed (Participants) | 70 | 91 | 93 | 93 | 97
  Anti-6B [Month 3] | 1.00 [0.73 to 1.38] | 0.94 [0.71 to 1.24] | 0.65 [0.50 to 0.86] | 1.06 [0.81 to 1.39] | 0.57 [0.45 to 0.73]
  Anti-6B [Month 9]: number analyzed (Participants) | 66 | 89 | 93 | 93 | 97
  Anti-6B [Month 9] | 2.26 [1.72 to 2.98] | 2.56 [2.01 to 3.25] | 2.05 [1.57 to 2.68] | 0.93 [0.75 to 1.15] | 1.98 [1.62 to 2.42]
  Anti-7F [Month 3] | 4.95 [3.82 to 6.41] | 3.69 [3.08 to 4.41] | 3.62 [3.12 to 4.19] | 4.77 [4.06 to 5.60] | 2.72 [2.30 to 3.22]
  Anti-7F [Month 9]: number analyzed (Participants) | 66 | 89 | 93 | 93 | 97
  Anti-7F [Month 9] | 9.92 [7.89 to 12.47] | 11.04 [9.29 to 13.11] | 8.98 [7.63 to 10.56] | 1.78 [1.49 to 2.13] | 6.47 [5.59 to 7.50]
  Anti-9V [Month 3] | 4.53 [3.39 to 6.05] | 4.25 [3.49 to 5.16] | 3.04 [2.51 to 3.69] | 5.13 [4.35 to 6.04] | 2.05 [1.61 to 2.61]
  Anti-9V [Month 9]: number analyzed (Participants) | 66 | 89 | 93 | 93 | 97
  Anti-9V [Month 9] | 10.09 [7.64 to 13.32] | 10.89 [9.11 to 13.03] | 9.55 [8.06 to 11.31] | 1.96 [1.58 to 2.43] | 6.51 [5.12 to 8.30]
  Anti-14 [Month 3]: number analyzed (Participants) | 70 | 91 | 93 | 93 | 97
  Anti-14 [Month 3] | 7.25 [5.37 to 9.81] | 6.77 [5.43 to 8.44] | 3.85 [3.18 to 4.68] | 5.27 [4.31 to 6.45] | 2.51 [1.98 to 3.19]
  Anti-14 [Month 9]: number analyzed (Participants) | 66 | 89 | 93 | 93 | 97
  Anti-14 [Month 9] | 11.50 [9.17 to 14.41] | 10.58 [8.60 to 13.00] | 7.33 [5.94 to 9.04] | 2.60 [2.01 to 3.37] | 5.08 [4.03 to 6.41]
  Anti-18C [Month 3]: number analyzed (Participants) | 69 | 91 | 93 | 94 | 97
  Anti-18C [Month 3] | 9.55 [7.19 to 12.67] | 9.48 [7.41 to 12.13] | 10.08 [8.25 to 12.31] | 13.20 [10.31 to 16.90] | 8.65 [6.44 to 11.60]
  Anti-18C [Month 9]: number analyzed (Participants) | 66 | 89 | 93 | 93 | 97
  Anti-18C [Month 9] | 20.26 [16.13 to 25.45] | 19.67 [15.89 to 24.35] | 25.47 [21.75 to 29.83] | 3.30 [2.55 to 4.27] | 32.29 [26.43 to 39.45]
  Anti-19F [Month 3]: number analyzed (Participants) | 70 | 91 | 93 | 93 | 97
  Anti-19F [Month 3] | 5.70 [4.06 to 8.02] | 11.15 [8.88 to 13.99] | 8.75 [7.37 to 10.38] | 10.93 [9.20 to 12.99] | 6.90 [5.62 to 8.48]
  Anti-19F [Month 9]: number analyzed (Participants) | 66 | 89 | 93 | 93 | 97
  Anti-19F [Month 9] | 8.00 [5.86 to 10.92] | 12.46 [10.47 to 14.84] | 8.88 [7.37 to 10.69] | 2.60 [2.03 to 3.31] | 9.47 [7.42 to 12.07]
  Anti-23F [Month 3]: number analyzed (Participants) | 70 | 91 | 93 | 93 | 97
  Anti-23F [Month 3] | 1.71 [1.23 to 2.37] | 1.52 [1.14 to 2.01] | 0.92 [0.72 to 1.19] | 1.59 [1.21 to 2.09] | 0.97 [0.74 to 1.27]
  Anti-23F [Month 9]: number analyzed (Participants) | 66 | 89 | 93 | 93 | 97
  Anti-23F [Month 9] | 4.00 [2.69 to 5.93] | 5.90 [4.37 to 7.96] | 3.83 [2.84 to 5.15] | 0.92 [0.68 to 1.23] | 3.40 [2.67 to 4.33]

3. Secondary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes.
Description: Concentrations were given in microgram per millilitre (µg/mL) and were expressed in geometric mean antibody concentrations. Pneumococcal vaccine serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Data were collected post-Dose 4 at Month 23 for the HIV+/+, HIV+/- and HIV- (3+1) groups and post-Dose 3 at Month 23 for HIV- (3+0) and HIV- (2+1) groups. The cut-off of the assay is 0.05 µg/mL.
Time Frame: up to study end at Month 23 (24-27 months of age)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 63 | 86 | 92 | 91 | 97
µg/mL
  Anti-1: number analyzed (Participants) | 63 | 86 | 92 | 90 | 97
  Anti-1 | 0.53 [0.35 to 0.80] | 0.74 [0.57 to 0.95] | 0.42 [0.34 to 0.53] | 0.28 [0.22 to 0.37] | 0.33 [0.26 to 0.41]
  Anti-4 | 0.56 [0.38 to 0.80] | 0.57 [0.46 to 0.71] | 0.44 [0.35 to 0.57] | 0.33 [0.25 to 0.44] | 0.34 [0.27 to 0.43]
  Anti-5: number analyzed (Participants) | 63 | 86 | 92 | 90 | 97
  Anti-5 | 0.79 [0.55 to 1.15] | 0.77 [0.61 to 0.97] | 0.72 [0.57 to 0.92] | 0.45 [0.36 to 0.57] | 0.52 [0.43 to 0.64]
  Anti-6B | 0.67 [0.42 to 1.06] | 0.73 [0.56 to 0.97] | 0.60 [0.47 to 0.77] | 0.76 [0.56 to 1.03] | 0.57 [0.44 to 0.74]
  Anti-7F | 1.25 [0.90 to 1.75] | 1.16 [0.96 to 1.39] | 1.08 [0.92 to 1.27] | 0.67 [0.54 to 0.83] | 0.84 [0.70 to 1.00]
  Anti-9V | 1.15 [0.77 to 1.71] | 1.30 [1.04 to 1.63] | 1.05 [0.86 to 1.28] | 0.85 [0.68 to 1.06] | 0.80 [0.64 to 1.00]
  Anti-14 | 2.62 [2.02 to 3.40] | 2.09 [1.69 to 2.58] | 1.32 [1.07 to 1.64] | 1.24 [0.96 to 1.61] | 1.06 [0.83 to 1.36]
  Anti-18C | 2.02 [1.41 to 2.89] | 1.60 [1.22 to 2.09] | 1.93 [1.58 to 2.35] | 0.80 [0.63 to 1.01] | 2.44 [1.97 to 3.02]
  Anti-19F | 2.01 [1.32 to 3.08] | 2.28 [1.72 to 3.02] | 2.53 [1.91 to 3.34] | 1.59 [1.15 to 2.20] | 2.22 [1.74 to 2.84]
  Anti-23F: number analyzed (Participants) | 63 | 86 | 92 | 90 | 97
  Anti-23F | 0.73 [0.49 to 1.09] | 0.85 [0.63 to 1.14] | 0.51 [0.39 to 0.67] | 0.53 [0.38 to 0.73] | 0.52 [0.37 to 0.72]

4. Secondary Outcome: Opsonophagocytic Titers Against Vaccine Pneumococcal Serotypes.
Description: Pneumococcal vaccine serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Data were collected post-Dose 3 at Month 3 and post-Dose 4 at Month 9 for the HIV+/+, HIV+/- and HIV- (3+1) groups,post-Dose 3 at Month 3 and at Month 9 for HIV- (3+0) group, and post-Dose 2 at Month 3 and post-Dose 3 at Month 9 for the HIV- (2+1) Group. Streptococcus pneumoniae opsonophagocytic activity was measured by a killing-assay using a HL 60 cell line. The results are presented as the dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions. The cut-off of the assay is an opsonic titer of 8.
Time Frame: At Month 3 and at Month 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 68 | 91 | 93 | 92 | 96
Titers
  Opsono-1 [Month 3] | 139.7 [85.2 to 229.0] | 147.6 [102.9 to 211.7] | 127.2 [86.2 to 187.8] | 268.7 [196.7 to 366.9] | 160.6 [117.8 to 218.8]
  Opsono-1 [Month 9]: number analyzed (Participants) | 63 | 85 | 90 | 89 | 94
  Opsono-1 [Month 9] | 1061.5 [680.5 to 1655.8] | 1377.8 [984.9 to 1927.4] | 1014.8 [768.4 to 1340.3] | 23.5 [16.1 to 34.4] | 1003.6 [763.2 to 1319.8]
  Opsono-4 [Month 3]: number analyzed (Participants) | 67 | 91 | 93 | 92 | 96
  Opsono-4 [Month 3] | 671.6 [430.7 to 1047.5] | 1518.1 [1149.7 to 2004.4] | 1711.9 [1367.7 to 2142.9] | 1890.6 [1547.2 to 2310.2] | 774.8 [596.7 to 1006.0]
  Opsono-4 [Month 9]: number analyzed (Participants) | 62 | 86 | 90 | 87 | 95
  Opsono-4 [Month 9] | 2034.2 [1593.5 to 2596.9] | 3259.0 [2579.2 to 4117.9] | 2484.7 [1919.0 to 3217.1] | 112.3 [70.8 to 178.1] | 1717.6 [1406.0 to 2098.2]
  Opsono-5 [Month 3] | 105.7 [73.8 to 151.4] | 128.6 [97.5 to 169.5] | 107.4 [81.8 to 141.0] | 189.2 [147.0 to 243.5] | 105.7 [81.6 to 136.8]
  Opsono-5 [Month 9]: number analyzed (Participants) | 63 | 85 | 90 | 90 | 94
  Opsono-5 [Month 9] | 540.4 [366.4 to 796.9] | 531.1 [397.3 to 710.0] | 630.2 [447.5 to 887.7] | 30.5 [21.8 to 42.5] | 472.7 [343.5 to 650.5]
  Opsono-6B [Month 3]: number analyzed (Participants) | 68 | 90 | 92 | 91 | 92
  Opsono-6B [Month 3] | 239.7 [123.0 to 467.4] | 480.5 [282.1 to 818.5] | 499.5 [286.1 to 872.2] | 1213.7 [808.2 to 1822.6] | 361.2 [221.8 to 588.2]
  Opsono-6B [Month 9]: number analyzed (Participants) | 60 | 84 | 88 | 86 | 94
  Opsono-6B [Month 9] | 853.0 [467.8 to 1555.3] | 986.6 [667.6 to 1457.9] | 1047.2 [679.3 to 1614.4] | 261.5 [161.0 to 424.7] | 945.9 [640.0 to 1398.2]
  Opsono-7F [Month 3]: number analyzed (Participants) | 68 | 90 | 92 | 92 | 95
  Opsono-7F [Month 3] | 4025.2 [2609.7 to 6208.4] | 10158.3 [7772.0 to 13277.2] | 5910.5 [4696.9 to 7437.6] | 6834.5 [5280.8 to 8845.4] | 2650.0 [2002.0 to 3507.9]
  Opsono-7F [Month 9]: number analyzed (Participants) | 63 | 85 | 88 | 90 | 95
  Opsono-7F [Month 9] | 10656.1 [7729.9 to 14690.0] | 18816.6 [14352.2 to 24669.7] | 12108.8 [9922.2 to 14777.4] | 2741.1 [2173.7 to 3456.5] | 6029.3 [4760.9 to 7635.6]
  Opsono-9V [Month 3]: number analyzed (Participants) | 68 | 90 | 93 | 92 | 96
  Opsono-9V [Month 3] | 1197.2 [796.2 to 1800.1] | 1736.5 [1224.1 to 2463.5] | 1672.2 [1243.6 to 2248.4] | 2216.0 [1760.9 to 2788.8] | 1068.2 [759.2 to 1503.0]
  Opsono-9V [Month 9]: number analyzed (Participants) | 64 | 86 | 91 | 90 | 94
  Opsono-9V [Month 9] | 2436.8 [1736.5 to 3419.7] | 3215.4 [2515.8 to 4109.6] | 4250.1 [3493.4 to 5170.8] | 492.3 [351.2 to 690.1] | 2572.5 [1890.3 to 3500.8]
  Opsono-14 [Month 3]: number analyzed (Participants) | 68 | 90 | 92 | 92 | 95
  Opsono-14 [Month 3] | 2656.2 [1686.7 to 4183.0] | 3175.1 [2472.8 to 4077.0] | 1902.7 [1300.9 to 2782.9] | 2205.0 [1648.8 to 2948.7] | 380.9 [228.1 to 636.0]
  Opsono-14 [Month 9]: number analyzed (Participants) | 65 | 87 | 89 | 87 | 94
  Opsono-14 [Month 9] | 2205.9 [1570.2 to 3099.0] | 2374.3 [1923.2 to 2931.2] | 2180.0 [1781.9 to 2667.0] | 280.0 [183.0 to 428.6] | 1152.9 [910.6 to 1459.6]
  Opsono-18C [Month 3]: number analyzed (Participants) | 68 | 91 | 91 | 92 | 93
  Opsono-18C [Month 3] | 438.7 [284.1 to 677.3] | 575.9 [442.9 to 748.8] | 1046.9 [802.6 to 1365.5] | 1203.2 [981.2 to 1475.4] | 1052.3 [777.7 to 1423.8]
  Opsono-18C [Month 9]: number analyzed (Participants) | 62 | 85 | 90 | 90 | 93
  Opsono-18C [Month 9] | 1039.3 [770.2 to 1402.3] | 1036.5 [800.1 to 1342.7] | 1344.4 [1074.6 to 1681.9] | 64.5 [44.1 to 94.3] | 1441.3 [1111.7 to 1868.5]
  Opsono-19F [Month 3]: number analyzed (Participants) | 68 | 91 | 92 | 92 | 95
  Opsono-19F [Month 3] | 228.6 [132.5 to 394.4] | 590.3 [418.9 to 831.6] | 511.9 [394.1 to 664.9] | 649.3 [481.1 to 876.2] | 275.9 [193.4 to 393.5]
  Opsono-19F [Month 9]: number analyzed (Participants) | 61 | 86 | 89 | 88 | 94
  Opsono-19F [Month 9] | 488.2 [275.3 to 865.9] | 1357.5 [976.2 to 1887.8] | 730.8 [516.5 to 1034.1] | 46.8 [31.6 to 69.5] | 630.3 [422.9 to 939.5]
  Opsono-23F [Month 3]: number analyzed (Participants) | 68 | 89 | 88 | 92 | 91
  Opsono-23F [Month 3] | 338.0 [174.1 to 656.2] | 769.6 [451.1 to 1312.9] | 864.1 [511.2 to 1460.6] | 1107.0 [683.0 to 1794.0] | 509.6 [306.8 to 846.6]
  Opsono-23F [Month 9]: number analyzed (Participants) | 63 | 87 | 90 | 86 | 95
  Opsono-23F [Month 9] | 1327.4 [736.2 to 2393.5] | 2120.7 [1359.4 to 3308.1] | 2144.8 [1312.5 to 3504.8] | 83.6 [47.2 to 148.0] | 1557.2 [1012.2 to 2395.7]

5. Secondary Outcome: Opsonophagocytic Titers Against Vaccine Pneumococcal Serotypes.
Description: Pneumococcal vaccine serotypes assessed were 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Data were collected post-Dose 4 at Month 23 for the HIV+/+, HIV+/- and HIV- (3+1) groups and post-Dose 3 at Month 23 for HIV- (3+0) and HIV- (2+1) groups. Streptococcus pneumoniae opsonophagocytic activity was measured by a killing-assay using a HL 60 cell line. The results are presented as the dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions. The cut-off of the assay is an opsonic titer of 8.
Time Frame: up to study end at Month 23 (24-27 months of age)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 59 | 84 | 89 | 86 | 91
Titers
  Opsono-1: number analyzed (Participants) | 59 | 84 | 89 | 85 | 91
  Opsono-1 | 36.7 [19.6 to 68.9] | 28.1 [17.4 to 45.4] | 22.8 [14.9 to 34.9] | 12.3 [8.2 to 18.6] | 13.9 [9.8 to 19.7]
  Opsono-4: number analyzed (Participants) | 53 | 74 | 82 | 79 | 83
  Opsono-4 | 76.6 [36.8 to 159.5] | 141.7 [79.2 to 253.5] | 125.5 [69.1 to 228.2] | 21.6 [12.4 to 37.5] | 58.8 [33.0 to 105.0]
  Opsono-5: number analyzed (Participants) | 57 | 82 | 88 | 86 | 89
  Opsono-5 | 22.5 [13.7 to 37.0] | 19.1 [13.9 to 26.2] | 19.5 [14.2 to 26.7] | 8.6 [6.5 to 11.3] | 13.3 [10.2 to 17.3]
  Opsono-6B: number analyzed (Participants) | 54 | 81 | 80 | 79 | 83
  Opsono-6B | 100.0 [48.8 to 204.7] | 75.5 [44.2 to 128.8] | 116.6 [63.7 to 213.3] | 87.2 [48.2 to 157.7] | 55.9 [32.0 to 97.7]
  Opsono-7F: number analyzed (Participants) | 55 | 80 | 81 | 77 | 81
  Opsono-7F | 6367.5 [4511.3 to 8987.6] | 7396.6 [5736.2 to 9537.6] | 6365.0 [5177.2 to 7825.4] | 5601.1 [4334.9 to 7237.3] | 5859.9 [4371.4 to 7855.2]
  Opsono-9V: number analyzed (Participants) | 53 | 80 | 85 | 84 | 89
  Opsono-9V | 507.6 [315.2 to 817.5] | 598.6 [396.9 to 902.7] | 1060.7 [761.2 to 1478.1] | 412.3 [267.4 to 635.9] | 465.7 [318.2 to 681.6]
  Opsono-14: number analyzed (Participants) | 56 | 79 | 84 | 76 | 80
  Opsono-14 | 452.0 [270.6 to 755.0] | 472.8 [305.1 to 732.6] | 362.3 [229.7 to 571.6] | 361.5 [213.2 to 613.2] | 185.2 [105.8 to 324.1]
  Opsono-18C: number analyzed (Participants) | 56 | 71 | 80 | 83 | 78
  Opsono-18C | 21.1 [13.0 to 34.4] | 26.7 [17.1 to 41.6] | 48.7 [30.4 to 78.1] | 9.8 [6.6 to 14.5] | 41.6 [27.3 to 63.3]
  Opsono-19F: number analyzed (Participants) | 55 | 74 | 86 | 82 | 85
  Opsono-19F | 41.8 [23.5 to 74.4] | 73.2 [47.0 to 114.0] | 52.5 [33.2 to 83.1] | 28.2 [17.8 to 44.6] | 47.6 [30.1 to 75.1]
  Opsono-23F: number analyzed (Participants) | 53 | 78 | 80 | 78 | 80
  Opsono-23F | 97.6 [38.2 to 249.6] | 154.8 [71.7 to 334.2] | 69.7 [31.7 to 153.1] | 92.7 [40.7 to 211.2] | 103.5 [47.0 to 227.7]

6. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A.
Description: Concentrations were given in microgram per millilitre (µg/mL) and were expressed in geometric mean antibody concentrations. Cross-reactive pneumococcal vaccine serotypes assessed were 6A and 19A. Data were collected post-Dose 3 at Month 3 and post-Dose 4 at Month 9 for the HIV+/+, HIV+/- and HIV- (3+1) groups,post-Dose 3 at Month 3 and at Month 9 for HIV- (3+0) group, and post-Dose 2 at Month 3 and post-Dose 3 at Month 9 for the HIV- (2+1) Group. The cut-off of the assay is 0.05 µg/mL.
Time Frame: At Month 3 and Month 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 70 | 91 | 93 | 93 | 97
µg/mL
  Anti-6A [Month 3] | 0.15 [0.12 to 0.19] | 0.12 [0.10 to 0.15] | 0.12 [0.10 to 0.15] | 0.13 [0.11 to 0.16] | 0.11 [0.09 to 0.13]
  Anti-6A [Month 9]: number analyzed (Participants) | 66 | 89 | 93 | 93 | 97
  Anti-6A [Month 9] | 0.48 [0.34 to 0.67] | 0.58 [0.43 to 0.77] | 0.36 [0.27 to 0.49] | 0.21 [0.15 to 0.28] | 0.36 [0.28 to 0.47]
  Anti-19A [Month 3]: number analyzed (Participants) | 69 | 91 | 93 | 92 | 97
  Anti-19A [Month 3] | 0.16 [0.12 to 0.23] | 0.28 [0.21 to 0.36] | 0.20 [0.16 to 0.25] | 0.29 [0.23 to 0.38] | 0.25 [0.20 to 0.32]
  Anti-19A [Month 9]: number analyzed (Participants) | 66 | 89 | 93 | 93 | 97
  Anti-19A [Month 9] | 0.99 [0.61 to 1.61] | 1.48 [1.06 to 2.08] | 0.78 [0.57 to 1.07] | 0.26 [0.19 to 0.37] | 1.04 [0.72 to 1.49]

7. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A.
Description: Concentrations were given in microgram per millilitre (µg/mL) and were expressed in geometric mean antibody concentrations. Cross-reactive pneumococcal vaccine serotypes assessed were 6A and 19A. Data were collected post-Dose 4 at Month 23 for the HIV+/+, HIV+/- and HIV- (3+1) groups and post-Dose 3 at Month 23 for HIV- (3+0) and HIV- (2+1) groups. The cut-off of the assay is 0.05 µg/mL.
Time Frame: up to study end at Month 23 (24-27 months of age)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 63 | 86 | 92 | 91 | 97
µg/mL
  Anti-6A | 0.23 [0.14 to 0.38] | 0.25 [0.17 to 0.35] | 0.20 [0.15 to 0.27] | 0.25 [0.18 to 0.36] | 0.19 [0.14 to 0.26]
  Anti-19A: number analyzed (Participants) | 63 | 86 | 92 | 89 | 97
  Anti-19A | 0.45 [0.26 to 0.76] | 0.47 [0.31 to 0.72] | 0.53 [0.35 to 0.80] | 0.41 [0.28 to 0.60] | 0.58 [0.41 to 0.83]

8. Secondary Outcome: Opsonophagocytic Titers Against Cross-reactive Pneumococcal Serotypes 6A and 19A.
Description: Cross-reactive pneumococcal vaccine serotypes assessed were 6A and 19A. Data were collected post-Dose 3 at Month 3 and post-Dose 4 at Month 9 for the HIV+/+, HIV+/- and HIV- (3+1) groups,post-Dose 3 at Month 3 and at Month 9 for HIV- (3+0) group, and post-Dose 2 at Month 3 and post-Dose 3 at Month 9 for the HIV- (2+1) Group. Streptococcus pneumoniae opsonophagocytic activity was measured by a killing-assay using a HL 60 cell line. The results are presented as the dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions. The cut-off of the assay is an opsonic titer of 8.
Time Frame: At Month 3 and at Month 9
Population: ATP cohort for immunogenicity included evaluable subjects for whom data concerning immunogenicity outcome measures were available. This included subjects for whom assay results were available for antibodies against at least 1 study vaccine antigen component post dose II or III, as applicable, or after booster vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 67 | 91 | 93 | 91 | 95
Titers
  Opsono -6A [Month 3]: number analyzed (Participants) | 67 | 91 | 89 | 91 | 95
  Opsono -6A [Month 3] | 7.7 [5.2 to 11.5] | 11.5 [7.4 to 17.9] | 12.1 [7.8 to 18.9] | 13.8 [9.1 to 20.9] | 8.1 [5.8 to 11.3]
  Opsono -6A [Month 9]: number analyzed (Participants) | 64 | 86 | 83 | 86 | 94
  Opsono -6A [Month 9] | 26.4 [14.7 to 47.3] | 38.6 [22.2 to 67.0] | 40.4 [22.9 to 71.4] | 9.5 [6.5 to 14.0] | 42.2 [25.5 to 69.9]
  Opsono -19A [Month 3]: number analyzed (Participants) | 66 | 91 | 93 | 90 | 95
  Opsono -19A [Month 3] | 9.5 [6.4 to 14.0] | 15.2 [10.4 to 22.2] | 10.6 [7.7 to 14.7] | 14.2 [9.7 to 20.8] | 7.8 [5.9 to 10.2]
  Opsono -19A [Month 9]: number analyzed (Participants) | 63 | 86 | 89 | 89 | 92
  Opsono -19A [Month 9] | 42.0 [24.8 to 71.2] | 101.8 [63.9 to 162.3] | 38.3 [24.1 to 60.9] | 7.9 [5.7 to 10.9] | 36.1 [22.3 to 58.3]

9. Secondary Outcome: Opsonophagocytic Titers Against Cross-reactive Pneumococcal Serotypes 6A and 19A.
Description: Cross-reactive pneumococcal vaccine serotypes assessed were 6A and 19A. Data were collected post-Dose 4 at Month 23 for the HIV+/+, HIV+/- and HIV- (3+1) groups and post-Dose 3 at Month 23 for HIV- (3+0) and HIV- (2+1) groups. Streptococcus pneumoniae opsonophagocytic activity was measured by a killing-assay using a HL 60 cell line. The results are presented as the dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions. The cut-off of the assay is an opsonic titer of 8.
Time Frame: up to study end at Month 23 (24-27 months of age)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 56 | 79 | 80 | 82 | 81
Titers
  Opsono-6A: number analyzed (Participants) | 53 | 79 | 79 | 79 | 79
  Opsono-6A | 14.2 [7.5 to 27.2] | 15.7 [9.4 to 26.2] | 20.5 [12.2 to 34.3] | 15.3 [8.5 to 27.5] | 19.0 [11.4 to 31.9]
  Opsono-19A | 19.9 [11.4 to 34.8] | 15.8 [10.0 to 24.8] | 25.1 [15.1 to 41.9] | 14.5 [9.4 to 22.6] | 16.8 [10.9 to 26.0]

10. Secondary Outcome: Concentrations of Antibodies Against Protein D (PD) by ELISA
Description: Concentrations of antibodies are presented as GMCs expressed as ELISA units per milliliter (EL.U/mL). The cut-off of the assay was 100 EL.U/mL. Data were collected post-Dose 3 at Month 3 and post-Dose 4 at Month 9 for the HIV+/+, HIV+/- and HIV- (3+1) groups,post-Dose 3 at Month 3 and at Month 9 for HIV- (3+0) group, and post-Dose 2 at Month 3 and post-Dose 3 at Month 9 for the HIV- (2+1) Group.
Time Frame: At Month 3 and at Month 9
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 70 | 91 | 93 | 94 | 97
EL.U/mL
  Anti-PD [Month 3] | 4215.1 [3622.3 to 4905.0] | 3397.6 [2917.2 to 3957.1] | 3431.8 [2955.1 to 3985.4] | 4253.1 [3721.0 to 4861.4] | 2240.0 [1871.0 to 2681.9]
  Anti-PD [Month 9]: number analyzed (Participants) | 66 | 89 | 93 | 93 | 97
  Anti-PD [Month 9] | 5443.1 [4705.0 to 6297.0] | 5018.3 [4335.7 to 5808.5] | 4576.5 [3938.2 to 5318.3] | 930.4 [770.0 to 1124.2] | 3141.0 [2619.0 to 3767.0]

11. Secondary Outcome: Concentrations of Antibodies Against Protein D (PD) by ELISA.
Description: Concentrations of antibodies are presented as GMCs expressed as ELISA units per milliliter (EL.U/mL). The cut-off of the assay was 100 EL.U/mL. Data were collected post-Dose 4 at Month 23 for the HIV+/+, HIV+/- and HIV- (3+1) groups and post-Dose 3 at Month 23 for HIV- (3+0) and HIV- (2+1) groups.
Time Frame: up to study end at Month 23 (24-27 months of age)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 63 | 86 | 92 | 91 | 97
EL.U/mL | 748.3 [581.8 to 962.3] | 615.3 [495.8 to 763.4] | 503.2 [421.0 to 601.5] | 421.3 [334.2 to 531.1] | 323.0 [255.6 to 408.1]

12. Secondary Outcome: Concentrations of Antibodies Against Diphtheria Toxoid (DT) and Tetanus Toxoid (TT).
Description: Concentrations of antibodies are presented as GMCs expressed as International units per millilitre (IU/mL) The cut-off of the assay is 0.1IU/mL.
Time Frame: 1 month following primary immunization (at Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 70 | 91 | 93 | 94 | 97
IU/mL
  Anti-DT: number analyzed (Participants) | 70 | 91 | 93 | 93 | 97
  Anti-DT | 2.42 [1.92 to 3.06] | 3.69 [3.19 to 4.26] | 3.42 [2.96 to 3.96] | 4.20 [3.76 to 4.68] | 3.00 [2.58 to 3.49]
  Anti-TT | 5.03 [4.16 to 6.07] | 4.77 [4.03 to 5.63] | 4.50 [3.89 to 5.21] | 5.03 [4.33 to 5.85] | 4.24 [3.50 to 5.14]

13. Secondary Outcome: Concentrations of Antibodies Against Diphtheria Toxoid (DT) and Tetanus Toxoid (TT).
Description: Concentrations of antibodies are presented as GMCs expressed as International units per millilitre (IU/mL). The cut-off of the assay is 0.1IU/mL.
Time Frame: 1 month after the booster dose of DTPw-HBV/Hib vaccine (at Month 15)
Population: The According-To-Protocol cohort for immunogenicity at 15-18 months included evaluable subjects from the ATP cohort for Immunogenicity who received the DTPw-HBV/Hib vaccine and for whom assay results were available for antibodies against at least 1 vaccine antigen component after this booster dose vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 59 | 81 | 91 | 87 | 92
IU/mL
  Anti-DT | 9.57 [7.91 to 11.59] | 11.70 [10.28 to 13.32] | 10.45 [9.18 to 11.89] | 12.67 [10.82 to 14.83] | 11.96 [10.48 to 13.64]
  Anti-TT | 14.44 [12.20 to 17.09] | 14.60 [12.58 to 16.95] | 16.19 [14.18 to 18.48] | 17.69 [15.57 to 20.11] | 19.77 [17.74 to 22.04]

14. Secondary Outcome: Concentrations of Antibodies Against Bordetella Pertussis (BPT) by ELISA.
Description: Concentrations of antibodies are presented as GMCs expressed as ELISA units per millilitre (EL.U/mL). The cut-off of the assay is 15 EL.U/mL.
Time Frame: 1 month following primary immunization (at Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 70 | 91 | 93 | 92 | 97
EL.U/mL | 90.86 [74.89 to 110.23] | 132.27 [118.60 to 147.51] | 143.08 [129.44 to 158.17] | 152.23 [137.86 to 168.10] | 146.60 [129.19 to 166.34]

15. Secondary Outcome: Concentrations of Antibodies Against Bordetella Pertussis (BPT) by ELISA .
Description: as for outcome 14
Time Frame: 1 month after the booster dose of DTPw-HBV/Hib vaccine (at Month 15)
Population: The ATP cohort for immunogenicityat 15-18 months included evaluable subjects from the ATP cohort for Immunogenicity who received the DTPw-HBV/Hib vaccine and for whom assay results were available for antibodies against at least 1 vaccine antigen component after this booster dose vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 59 | 81 | 90 | 87 | 92
EL.U/mL | 161.01 [131.88 to 196.58] | 227.01 [202.86 to 254.03] | 241.77 [218.18 to 267.90] | 259.45 [234.70 to 286.81] | 267.80 [243.49 to 294.54]

16. Secondary Outcome: Concentrations of Antibodies Against Polyribosyl-ribitol Phosphate (PRP)
Description: Concentrations of antibodies are presented as GMCs expressed as microgram per millilitre (µg/mL). The cut-off of the assay is 0.15 µg/mL.
Time Frame: 1 month following primary immunization (at Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 70 | 91 | 93 | 93 | 97
µg/mL | 16.71 [11.63 to 24.01] | 20.55 [15.78 to 26.78] | 20.36 [15.56 to 26.64] | 24.22 [18.45 to 31.80] | 21.78 [16.47 to 28.79]

17. Secondary Outcome: Concentrations of Antibodies Against Polyribosyl-ribitol Phosphate (PRP)
Description: as for outcome 16
Time Frame: 1 month after the booster vaccination (at Month 15)
Population: The ATP cohort for immunogenicity at 15 -18 months included evaluable subjects from the ATP cohort for Immunogenicity who received the DTPw-HBV/Hib vaccine and for whom assay results were available for antibodies against at least 1 vaccine antigen component after this booster dose vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 59 | 80 | 91 | 87 | 92
µg/mL | 50.11 [33.29 to 75.43] | 71.23 [55.03 to 92.19] | 83.46 [64.51 to 107.98] | 93.18 [69.67 to 124.64] | 129.99 [103.73 to 162.89]

18. Secondary Outcome: Concentrations of Antibodies Against Hepatitis B Surface Antigen (HBs) by ELISA
Description: Concentrations of antibodies are presented as GMCs expressed as milli-International units per milliliter (mIU/mL). The cut-off of the assay is 10 mIU/mL.
  As a decrease in the specificity of the anti-HBs ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL), the table showed results following partial or complete retesting/reanalysis
Time Frame: 1 month following primary immunization (at Month 3)
Population: According-To-Protocol cohort for immunogenicity included evaluable subjects for whom data concerning immunogenicity outcome measures were available. This included subjects for whom assay results were available for antibodies against at least 1 study vaccine antigen component post dose II or III, as applicable, or after booster vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 63 | 85 | 88 | 87 | 90
mIU/mL | 288.45 [167.12 to 497.86] | 478.53 [333.22 to 687.22] | 865.5 [654.8 to 1144.1] | 904.7 [646.0 to 1267.0] | 563.5 [373.8 to 849.4]

19. Secondary Outcome: Concentrations of Antibodies Against Hepatitis B Surface Antigen (HBs) by ELISA.
Description: Concentrations of antibodies were presented as GMCs expressed as milli-International units per milliliter (mIU/mL). The cut-off of the assay was 10 mIU/mL.
  As a decrease in the specificity of the anti-HBs ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL), the table showed results following partial or complete retesting/reanalysis
Time Frame: 1 month after the booster dose of DTPw-HBV/Hib vaccine (at Month 15)
Population: The ATP cohort for immunogenicity at 15-18 months included evaluable subjects from the ATP cohort for Immunogenicity who received the DTPw-HBV/Hib vaccine and for whom assay results were available for antibodies against at least 1 vaccine antigen component after this booster dose vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 58 | 78 | 90 | 81 | 89
mIU/mL | 1871.0 [892.9 to 3920.7] | 2507.4 [1500.7 to 4189.4] | 3674.4 [2446.9 to 5517.9] | 4287.6 [2785.9 to 6598.8] | 3583.4 [2194.8 to 5850.6]

20. Secondary Outcome: Concentrations of Antibodies Against Rotavirus Immunoglobulin A (Rotavirus IgA), by Rotarix Vaccination Status.
Description: Concentrations of antibodies are presented as GMCs expressed as units per millilitre (U/mL). The cut-off of the assay is 20 U/mL. Data were collected for subjects who received 1, 2 doses or no Rotarix dose during the study.
Time Frame: 1 month after the administration of the second vaccine dose (at Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 58 | 59 | 66 | 66 | 67
U/mL
  Anti-rotavirus IgA [1 dose]: number analyzed (Participants) | 58 | 59 | 1 | 1 | 67
  Anti-rotavirus IgA [1 dose] | NA [NA to NA] — No subject in this group received 1 dose of Rotarix. | NA [NA to NA] — No subject in this group received 1 dose of Rotarix. | 25.0 [NA to NA] — Not calculable because of too few subjects | NA [NA to NA] — Values were below the assay cut-off value of 20 U/mL | NA [NA to NA] — No subject in this group received 1 dose of Rotarix.
  Anti-rotavirus IgA [2 doses] | 52.6 [33.8 to 81.8] | 104.1 [66.3 to 163.5] | 146.4 [94.2 to 227.4] | 92.0 [60.0 to 141.0] | 74.3 [47.5 to 116.3]
  Anti-rotavirus IgA [0 dose]: number analyzed (Participants) | 11 | 27 | 25 | 24 | 28
  Anti-rotavirus IgA [0 dose] | 54.8 [13.1 to 229.2] | 54.0 [21.3 to 136.8] | 63.1 [34.8 to 114.5] | 47.5 [26.5 to 85.3] | 41.7 [22.3 to 78.1]

21. Secondary Outcome: Concentrations of Antibodies Against Measles
Description: Concentrations of antibodies are presented as GMCs expressed as milli-International units per milliliter (mIU/mL).The cut-off of the assay is 150 mIU/mL.
Time Frame: 1 month following administration of the 1st and 2nd vaccine dose (at Months 9 and 15)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 63 | 85 | 91 | 87 | 93
mIU/mL
  Anti-Measles [Month 9]: number analyzed (Participants) | 54 | 79 | 82 | 83 | 87
  Anti-Measles [Month 9] | 2013.36 [1566.36 to 2587.94] | 1917.14 [1468.59 to 2502.68] | 1973.84 [1512.90 to 2575.22] | 1509.36 [1157.32 to 1968.50] | 1719.76 [1360.39 to 2174.08]
  Anti-Measles [Month 15] | 3358.15 [2578.34 to 4373.83] | 4189.83 [3451.63 to 5085.91] | 3713.51 [3050.30 to 4520.92] | 3311.30 [2698.56 to 4063.17] | 3204.79 [2659.00 to 3862.61]

22. Secondary Outcome: Anti-LytC IgA and Anti-PhtD IgA Antibodies Concentrations in Salivary Samples
Description: Salivary antibodies against selected common bacterial protein antigens. Salivary samples (1.0 mL) were collected by using an Oracol™ device consisting of a sponge (2 cm3) placed on a stick that was used to brush the teeth and gums to absorb the saliva. Salivary samples were sent to RMPRU (or GSK Biologicals' designated validated laboratory) where the sponge was centrifuged to extract the saliva and that was immediately stored at -70°C. The cut-off of the assay was 2.3 U/mL for anti-LytC IgA and 2.2 U/mL for anti PhtD IgA.
Time Frame: up to study end at Month 23 (24-27 months of age)
Population: The Total Vaccinated cohort included all subjects with at least one vaccine dose administration documented
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 77 | 95 | 98 | 94 | 98
U/mL
  Anti-LytC [Month0]: number analyzed (Participants) | 65 | 50 | 46 | 46 | 45
  Anti-LytC [Month0] | 7.71 [5.44 to 10.95] | 5.49 [3.81 to 7.91] | 6.22 [4.35 to 8.90] | 5.98 [4.24 to 8.43] | 6.67 [4.89 to 9.08]
  Anti-LytC [Month3]: number analyzed (Participants) | 74 | 79 | 95 | 91 | 93
  Anti-LytC [Month3] | 18.30 [13.29 to 25.22] | 13.48 [10.46 to 17.37] | 13.29 [10.50 to 16.82] | 13.81 [10.56 to 18.06] | 14.43 [11.32 to 18.39]
  Anti-LytC [Month8]: number analyzed (Participants) | 75 | 95 | 98 | 94 | 98
  Anti-LytC [Month8] | 27.23 [18.88 to 39.29] | 15.99 [12.29 to 20.79] | 24.51 [18.63 to 32.24] | 22.64 [16.56 to 30.96] | 21.85 [16.32 to 29.25]
  Anti-LytC [Month9]: number analyzed (Participants) | 77 | 94 | 98 | 94 | 97
  Anti-LytC [Month9] | 30.96 [20.88 to 45.88] | 15.54 [11.72 to 20.61] | 24.60 [17.89 to 33.83] | 21.06 [15.15 to 29.27] | 25.00 [18.66 to 33.50]
  Anti-LytC [Month11]: number analyzed (Participants) | 77 | 93 | 98 | 93 | 97
  Anti-LytC [Month11] | 37.01 [24.64 to 55.59] | 18.79 [13.94 to 25.32] | 43.03 [30.64 to 60.44] | 35.65 [26.47 to 48.02] | 38.07 [28.23 to 51.34]
  Anti-LytC [Month14]: number analyzed (Participants) | 73 | 94 | 98 | 94 | 97
  Anti-LytC [Month14] | 39.45 [28.22 to 55.15] | 24.69 [18.48 to 32.97] | 39.59 [28.87 to 54.29] | 38.87 [29.26 to 51.63] | 34.75 [26.40 to 45.74]
  Anti-LytC [Month15]: number analyzed (Participants) | 74 | 93 | 97 | 93 | 98
  Anti-LytC [Month15] | 58.11 [38.95 to 86.69] | 28.09 [21.12 to 37.36] | 42.43 [31.21 to 57.68] | 50.45 [38.70 to 65.77] | 42.98 [32.28 to 57.22]
  Anti-LytC [Month23]: number analyzed (Participants) | 73 | 91 | 97 | 92 | 98
  Anti-LytC [Month23] | 89.32 [63.92 to 124.81] | 43.61 [32.16 to 59.14] | 68.34 [51.15 to 91.32] | 61.40 [48.68 to 77.45] | 59.75 [45.69 to 78.12]
  Anti-PhtD [Month0]: number analyzed (Participants) | 65 | 50 | 46 | 46 | 45
  Anti-PhtD [Month0] | 4.58 [3.36 to 6.25] | 3.83 [2.83 to 5.18] | 7.85 [5.18 to 11.90] | 6.30 [4.39 to 9.04] | 5.49 [3.73 to 8.08]
  Anti-PhtD [Month3]: number analyzed (Participants) | 74 | 79 | 95 | 91 | 93
  Anti-PhtD [Month3] | 5.49 [3.97 to 7.59] | 4.92 [3.75 to 6.45] | 5.14 [4.07 to 6.49] | 5.06 [3.96 to 6.47] | 5.10 [4.02 to 6.47]
  Anti-PhtD [Month8]: number analyzed (Participants) | 75 | 95 | 98 | 94 | 98
  Anti-PhtD [Month8] | 7.77 [5.46 to 11.06] | 5.86 [4.51 to 7.62] | 9.49 [7.10 to 12.69] | 10.01 [7.10 to 14.12] | 8.35 [6.22 to 11.21]
  Anti-PhtD [Month9]: number analyzed (Participants) | 77 | 94 | 98 | 94 | 97
  Anti-PhtD [Month9] | 9.16 [6.37 to 13.17] | 7.32 [5.50 to 9.73] | 16.47 [11.34 to 23.94] | 14.01 [9.77 to 20.11] | 11.71 [8.45 to 16.23]
  Anti-PhtD [Month11]: number analyzed (Participants) | 77 | 93 | 98 | 93 | 97
  Anti-PhtD [Month11] | 9.49 [6.86 to 13.14] | 7.92 [5.76 to 10.90] | 16.93 [11.58 to 24.75] | 15.41 [10.83 to 21.94] | 15.70 [11.36 to 21.70]
  Anti-PhtD [Month14]: number analyzed (Participants) | 73 | 94 | 98 | 94 | 97
  Anti-PhtD [Month14] | 14.06 [9.92 to 19.92] | 10.74 [8.01 to 14.40] | 19.39 [13.98 to 26.87] | 22.04 [16.09 to 30.20] | 14.54 [10.62 to 19.92]
  Anti-PhtD [Month15]: number analyzed (Participants) | 74 | 93 | 98 | 93 | 98
  Anti-PhtD [Month15] | 15.04 [10.08 to 22.46] | 11.35 [8.27 to 15.59] | 18.06 [13.04 to 25.02] | 24.03 [17.55 to 32.92] | 17.07 [12.08 to 24.12]
  Anti-PhtD [Month23]: number analyzed (Participants) | 73 | 91 | 97 | 92 | 98
  Anti-PhtD [Month23] | 41.41 [27.82 to 61.62] | 29.17 [20.84 to 40.83] | 39.84 [28.47 to 55.75] | 35.69 [26.26 to 48.50] | 35.92 [26.60 to 48.52]

23. Secondary Outcome: Number of Swabs With Positive Cultures of Haemophilus Influenzae and/or Streptococcus Pneumoniae (Vaccine Serotypes, Cross-reactive or Other Serotypes) and Other Bacterial Pathogens in the Nasopharynx.
Description: Positive cultures of H. influenza* (HI) and S. pneumonia(SP) and other bacterial pathogens such as Moraxella catarrhalis(MC), Group A streptococci and Staphylococcus aureus (SA), identified in the nasopharynx at each swab time point: Month (Mth) 0 (Pre-vaccination time point at 6-12 weeks of age), Mth 3 (18 weeks of age), Mth 8 (9-10 Months of age), Mth 9 (10-11 Months of age), Mth 11 (12-13 Months of age), Mth 14 (15-18 Months of age), Mth 15 (16-19 Months of age) and Mth 23 (24-27 Months of age). *Data presented included only results from samples confirmed as positive for Hi/Non Typeable Hi after differentiation from H. haemolyticus by Polymerase Chain Reaction (PCR) assay
Time Frame: up to study end at Month 23 (24-27 months of age)
Population: The Total Vaccinated cohort included all subjects with at least one vaccine dose administration documented
Measure: Number; unit: Swabs
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 83 | 101 | 100 | 100 | 100
Swabs
  Any SP - Mth 0 | 23 | 24 | 25 | 30 | 17
  Any SP - Mth 3: number analyzed (Participants) | 81 | 98 | 98 | 95 | 98
  Any SP - Mth 3 | 47 | 62 | 58 | 55 | 64
  Any SP - Mth 8: number analyzed (Participants) | 76 | 95 | 98 | 94 | 98
  Any SP - Mth 8 | 55 | 61 | 65 | 67 | 67
  Any SP - Mth 9: number analyzed (Participants) | 77 | 96 | 98 | 94 | 98
  Any SP - Mth 9 | 50 | 64 | 62 | 66 | 70
  Any SP - Mth 11: number analyzed (Participants) | 77 | 94 | 98 | 94 | 97
  Any SP - Mth 11 | 52 | 61 | 67 | 62 | 70
  Any SP - Mth 14: number analyzed (Participants) | 75 | 94 | 98 | 94 | 98
  Any SP - Mth 14 | 52 | 64 | 69 | 70 | 70
  Any SP - Mth 15: number analyzed (Participants) | 75 | 94 | 98 | 94 | 98
  Any SP - Mth 15 | 59 | 68 | 62 | 70 | 68
  Any SP - Mth 23: number analyzed (Participants) | 73 | 92 | 97 | 92 | 98
  Any SP - Mth 23 | 58 | 59 | 63 | 60 | 66
  Any HI - Mth 0: number analyzed (Participants) | 82 | 101 | 99 | 100 | 98
  Any HI - Mth 0 | 14 | 12 | 17 | 12 | 12
  Any HI - Mth 3: number analyzed (Participants) | 80 | 98 | 98 | 95 | 98
  Any HI - Mth 3 | 30 | 34 | 36 | 33 | 37
  Any HI - Mth 8: number analyzed (Participants) | 77 | 94 | 97 | 94 | 98
  Any HI - Mth 8 | 21 | 41 | 34 | 30 | 38
  Any HI - Mth 9: number analyzed (Participants) | 77 | 96 | 97 | 94 | 98
  Any HI - Mth 9 | 28 | 47 | 34 | 29 | 32
  Any HI - Mth 11: number analyzed (Participants) | 76 | 93 | 96 | 88 | 92
  Any HI - Mth 11 | 33 | 44 | 36 | 34 | 40
  Any HI - Mth 14: number analyzed (Participants) | 68 | 81 | 81 | 73 | 82
  Any HI - Mth 14 | 29 | 39 | 38 | 31 | 27
  Any HI - Mth 15: number analyzed (Participants) | 75 | 94 | 98 | 94 | 98
  Any HI - Mth 15 | 35 | 54 | 54 | 51 | 55
  Any HI - Mth 23: number analyzed (Participants) | 73 | 92 | 97 | 92 | 98
  Any HI - Mth 23 | 39 | 45 | 58 | 53 | 62
  Any MC - Mth 0 | 35 | 39 | 42 | 42 | 44
  Any MC - Mth 3: number analyzed (Participants) | 81 | 98 | 98 | 95 | 98
  Any MC - Mth 3 | 63 | 88 | 88 | 87 | 90
  Any MC - Mth 8: number analyzed (Participants) | 77 | 95 | 98 | 94 | 98
  Any MC - Mth 8 | 56 | 83 | 84 | 79 | 82
  Any MC - Mth 9: number analyzed (Participants) | 77 | 96 | 98 | 94 | 98
  Any MC - Mth 9 | 62 | 79 | 75 | 81 | 72
  Any MC - Mth 11: number analyzed (Participants) | 77 | 94 | 98 | 94 | 97
  Any MC - Mth 11 | 69 | 80 | 73 | 73 | 83
  Any MC - Mth 14: number analyzed (Participants) | 75 | 94 | 98 | 94 | 98
  Any MC - Mth 14 | 65 | 81 | 84 | 90 | 84
  Any MC - Mth 15: number analyzed (Participants) | 75 | 94 | 98 | 94 | 98
  Any MC - Mth 15 | 60 | 82 | 83 | 87 | 86
  Any MC - Mth 23: number analyzed (Participants) | 73 | 92 | 97 | 92 | 98
  Any MC - Mth 23 | 59 | 73 | 78 | 71 | 79
  Any SA - Mth 0 | 37 | 48 | 56 | 57 | 55
  Any SA - Mth 3: number analyzed (Participants) | 81 | 98 | 98 | 95 | 98
  Any SA - Mth 3 | 41 | 37 | 37 | 40 | 32
  Any SA - Mth 11: number analyzed (Participants) | 77 | 94 | 98 | 94 | 97
  Any SA - Mth 11 | 9 | 18 | 13 | 13 | 19
  Any SA - Mth 8: number analyzed (Participants) | 77 | 95 | 98 | 94 | 98
  Any SA - Mth 8 | 16 | 18 | 13 | 19 | 24
  Any SA - Mth 9: number analyzed (Participants) | 77 | 96 | 98 | 94 | 98
  Any SA - Mth 9 | 19 | 26 | 18 | 16 | 17
  Any SA - Mth 14: number analyzed (Participants) | 75 | 94 | 98 | 94 | 98
  Any SA - Mth 14 | 11 | 15 | 9 | 13 | 13
  Any SA - Mth 15: number analyzed (Participants) | 75 | 94 | 98 | 94 | 98
  Any SA - Mth 15 | 12 | 11 | 20 | 13 | 18
  Any SA - Mth 23: number analyzed (Participants) | 73 | 92 | 97 | 92 | 98
  Any SA - Mth 23 | 8 | 16 | 10 | 13 | 18

24. Secondary Outcome: Number of Subjects With Acquisition of New Streptococcus Pneumoniae and Haemophilus Influenzae Strains Identified in Nasopharyngeal Swabs
Description: Acquisition of new H. influenza* (HI) and S. pneumonia(SP) strains, identified in the nasopharynx at each swab time point: Month (Mth) 3 (18 weeks of age), Mth 8 (9-10 Months of age), Mth 9 (10-11 Months of age), Mth 11 (12-13 Months of age), Mth 14 (15-18 Months of age), Mth 15 (16-19 Months of age) and Mth 23 (24-27 Months of age). *Data presented included only results from samples confirmed as positive for Hi/Non Typeable Hi after differentiation from H. haemolyticus by PCR assay
Time Frame: up to study end at Month 23 (24-27 months of age)
Population: The Total Vaccinated cohort included all subjects with at least one vaccine dose administration documented
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 81 | 98 | 98 | 95 | 98
Participants
  Any SP - Mth 3 | 35 | 47 | 46 | 41 | 56
  Any SP - Mth 8: number analyzed (Participants) | 77 | 95 | 98 | 94 | 98
  Any SP - Mth 8 | 59 | 68 | 70 | 67 | 76
  Any SP - Mth 9: number analyzed (Participants) | 77 | 95 | 98 | 94 | 98
  Any SP - Mth 9 | 64 | 76 | 77 | 78 | 82
  Any SP - Mth 11: number analyzed (Participants) | 77 | 93 | 98 | 94 | 97
  Any SP - Mth 11 | 69 | 79 | 84 | 84 | 90
  Any SP - Mth 14: number analyzed (Participants) | 75 | 92 | 98 | 94 | 97
  Any SP - Mth 14 | 68 | 82 | 90 | 90 | 93
  Any SP - Mth 15: number analyzed (Participants) | 75 | 92 | 98 | 94 | 97
  Any SP - Mth 15 | 72 | 86 | 90 | 92 | 94
  Any SP - Mth 23: number analyzed (Participants) | 73 | 90 | 97 | 92 | 97
  Any SP - Mth 23 | 72 | 87 | 95 | 90 | 96
  Any HI - Mth 3: number analyzed (Participants) | 80 | 98 | 97 | 95 | 96
  Any HI - Mth 3 | 26 | 25 | 27 | 29 | 30
  Any HI - Mth 8: number analyzed (Participants) | 76 | 94 | 96 | 94 | 96
  Any HI - Mth 8 | 34 | 49 | 48 | 42 | 45
  Any HI - Mth 9: number analyzed (Participants) | 76 | 94 | 95 | 94 | 96
  Any HI - Mth 9 | 45 | 63 | 52 | 52 | 57
  Any HI - Mth 11: number analyzed (Participants) | 75 | 91 | 94 | 88 | 92
  Any HI - Mth 11 | 55 | 67 | 60 | 57 | 65
  Any HI - Mth 14: number analyzed (Participants) | 67 | 78 | 78 | 70 | 78
  Any HI - Mth 14 | 56 | 60 | 58 | 54 | 59
  Any HI - Mth 15: number analyzed (Participants) | 67 | 78 | 78 | 70 | 70
  Any HI - Mth 15 | 59 | 67 | 64 | 58 | 65
  Any HI - Mth 23: number analyzed (Participants) | 65 | 76 | 77 | 69 | 78
  Any HI - Mth 23 | 60 | 70 | 71 | 59 | 71

25. Secondary Outcome: Number of Subjects With Any and Severe (Grade 3) Solicited Local Adverse Events (AEs).
Description: Solicited local AEs assessed were pain, redness and swelling. Any = incidence of any local symptom regardless of intensity grade. Grade 3 pain = cried when limb was moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling above 30 millimetre.
Time Frame: During the 4-day (Days 0-3) post-primary vaccination period across doses
Population: The Total Vaccinated cohort included all subjects who received at least one vaccine dose administration, with analysis done solely on subjects for whom post-vaccination results about solicited symptoms were available.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 83 | 101 | 98 | 98 | 98
Participants
  Any pain | 73 | 93 | 92 | 95 | 97
  Grade 3 pain | 18 | 18 | 28 | 42 | 34
  Any redness | 62 | 80 | 83 | 83 | 84
  Redness > 30 mm | 14 | 10 | 17 | 20 | 14
  Any swelling | 67 | 83 | 84 | 91 | 84
  Swelling > 30 mm | 23 | 32 | 41 | 44 | 31

26. Secondary Outcome: Number of Subjects With Any, Severe (Grade 3) and Related Solicited General Adverse Events (AEs).
Description: General AEs = diarrhoea, drowsiness, irritability, loss of appetite, vomiting and fever (axillary ≥ 37.5 degrees Celsius). Any= Incidence of any symptom regardless of intensity grade or relationship to vaccination. Grade 3:
  drowsiness = prevented normal activity. irritability = crying that could not be comforted/ prevented normal activity. loss of appetite = not eating at all. diarrhoea: ≥ 6 looser than normal stools/day. vomiting: ≥ 3 episodes of vomiting/day. Fever = > 39.5°C Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Days 0-3) post-primary vaccination period across doses
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 83 | 101 | 98 | 98 | 98
Participants
  Any diarrhoea | 8 | 5 | 12 | 10 | 5
  Grade 3 diarrhoea | 2 | 0 | 3 | 3 | 2
  Related diarrhoea | 8 | 5 | 11 | 9 | 5
  Any drowsiness | 49 | 62 | 70 | 70 | 68
  Grade 3 drowsiness | 1 | 6 | 5 | 7 | 8
  Related drowsiness | 47 | 58 | 67 | 66 | 63
  Fever (axillary) >= 37.5°C | 38 | 36 | 41 | 28 | 28
  Fever (axillary) > 39.5°C | 0 | 0 | 2 | 0 | 0
  Related fever | 33 | 30 | 38 | 27 | 25
  Any irritability | 63 | 84 | 89 | 89 | 91
  Grade 3 irritability | 6 | 10 | 19 | 13 | 15
  Related irritability | 62 | 80 | 86 | 83 | 85
  Any loss of appetite | 36 | 53 | 56 | 57 | 62
  Grade 3 loss of appetite | 0 | 1 | 2 | 2 | 5
  Related loss of appetite | 35 | 47 | 53 | 53 | 58
  Any vomiting | 17 | 19 | 15 | 18 | 23
  Grade 3 vomiting | 3 | 3 | 4 | 5 | 2
  Related vomiting | 16 | 16 | 14 | 13 | 17

27. Secondary Outcome: Number of Subjects With Any and Severe (Grade 3) Solicited Local Adverse Events (AEs).
Description: as for outcome 25
Time Frame: During the 4-day (Days 0-3) period following booster vaccination with Synflorix vaccine
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 74 | 95 | 96 | 0 | 96
Participants
  Any pain | 40 | 58 | 62 |  | 60
  Grade 3 pain | 2 | 1 | 2 |  | 6
  Any redness | 25 | 31 | 39 |  | 45
  Redness > 30 mm | 5 | 1 | 3 |  | 0
  Any swelling | 28 | 39 | 38 |  | 53
  Swelling > 30 mm | 5 | 4 | 8 |  | 10

28. Secondary Outcome: Number of Subjects With Any, Severe (Grade 3) and Related Solicited General Adverse Events (AEs).
Description: Solicited general AEs = drowsiness, irritability, loss of appetite and fever (axillary ≥ 37.5 degrees Celsius). Any= Incidence of any symptom regardless of intensity grade or relationship to vaccination. Grade 3:
  drowsiness = prevented normal activity. irritability = crying that could not be comforted/ prevented normal activity. loss of appetite = not eating at all. Fever = temperature > 39.5°C Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 4-day (Days 0-3) period following booster vaccination with Synflorix vaccine
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 74 | 95 | 96 | 0 | 96
Participants
  Any drowsiness | 17 | 28 | 34 |  | 33
  Grade 3 drowsiness | 2 | 0 | 1 |  | 1
  Related drowsiness | 16 | 27 | 31 |  | 32
  Fever >= 37.5°C | 9 | 11 | 7 |  | 11
  Fever > 39.5°C | 0 | 0 | 0 |  | 0
  Related fever | 8 | 10 | 7 |  | 10
  Any irritability | 25 | 35 | 31 |  | 43
  Grade 3 irritability | 4 | 1 | 1 |  | 1
  Related irritability | 24 | 35 | 31 |  | 42
  Any loss of appetite | 17 | 23 | 29 |  | 37
  Grade 3 loss of appetite | 0 | 0 | 1 |  | 2
  Related loss of appetite | 16 | 23 | 29 |  | 33

29. Secondary Outcome: Number of Subjects With Unsolicited AEs.
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within the 31-day (Days 0-30) post-primary vaccination period
Population: The Total Vaccinated cohort included all subjects with at least one vaccine dose administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 83 | 101 | 100 | 100 | 100
Participants | 73 | 92 | 93 | 90 | 97

30. Secondary Outcome: Number of Subjects With Unsolicited AEs.
Description: as for outcome 29
Time Frame: Within the 31-day (Days 0-30) post Synflorix booster vaccination period
Population: The Total Vaccinated cohort included all subjects with at least one vaccine dose administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 76 | 96 | 98 | 0 | 98
Participants | 35 | 47 | 50 |  | 44

31. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: From study start at Month 0 (6 weeks of age and above) up to study end at Month 23 (24-27 months of age)
Population: The Total Vaccinated cohort included all subjects with at least one vaccine dose administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Number analyzed (Participants) | 83 | 101 | 100 | 100 | 100
Participants | 31 | 25 | 20 | 15 | 20

ADVERSE EVENTS:
Time Frame: SAEs: from Month 0 up to Month 23. Unsolicited AEs: within the 31-day post-primary and post Synflorix booster vaccination period. Solicited AEs: During the 4-day period following the primary and the Synflorix booster vaccination.
Arm/Group | HIV+/+ Group | HIV+/- Group | HIV- (3+1) Group | HIV- (3+0) Group | HIV- (2+1) Group
Serious Adverse Events (participants affected / at risk) | 31/83 | 25/101 | 20/100 | 15/100 | 20/100
Other Adverse Events (participants affected / at risk) | 83/83 | 100/101 | 98/100 | 98/100 | 98/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV+/+ Group (N=83) | HIV+/- Group (N=101) | HIV- (3+1) Group (N=100) | HIV- (3+0) Group (N=100) | HIV- (2+1) Group (N=100)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Cerebral palsy (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Trisomy 21 (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Ventricular septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Death (General disorders) | 1 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 2 | 0 | 0 | 1 | 0
Sudden infant death syndrome (General disorders) | 0 | 1 | 0 | 0 | 0
Hepatitis neonatal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0 | 0
AIDS dementia complex (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 1 | 3 | 4 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 13 | 5 | 6 | 1 | 8
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 8 | 8 | 5 | 4 | 4
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1 | 0 | 0 | 0
H1N1 influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0
HIV infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Injection site abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Measles (Infections and infestations) | 1 | 2 | 0 | 1 | 1
Meningitis meningococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Meningitis tuberculous (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 4 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 3 | 0 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 11 | 1 | 1 | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Subacute endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2
Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 3 | 1 | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Electric shock (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Herbal toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Near drowning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Kwashiorkor (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 0
Marasmus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0 | 2 | 0
Encephalitis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 1 | 3 | 1 | 2
Renal impairment (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | HIV+/+ Group (N=83) | HIV+/- Group (N=101) | HIV- (3+1) Group (N=100) | HIV- (3+0) Group (N=100) | HIV- (2+1) Group (N=100)
Diarrhoea (Gastrointestinal disorders) | 13 | 16 | 18 | 13 | 11 — Within the 31-day (Days 0-30) post-primary vaccination period
Diarrhoea (Gastrointestinal disorders) | 5/76 | 10/96 | 10/98 | 0/0 | 8/98 — Within the 31-day (Days 0-30) post Synflorix booster vaccination period
Vomiting (Gastrointestinal disorders) | 18 | 16 | 11 | 15 | 12 — Within the 31-day (Days 0-30) post-primary vaccination period
Vomiting (Gastrointestinal disorders) | 1/76 | 8/96 | 7/98 | 0/0 | 5/98 — Within the 31-day (Days 0-30) post Synflorix booster vaccination period
Diarrhoea (General disorders) | 8 | 5 | 12/98 | 10/98 | 5/98 — During the 4-day (Days 0-3) post-primary vaccination period
Drowsiness (General disorders) | 49 | 62 | 70/98 | 70/98 | 68/98 — During the 4-day (Days 0-3) post-primary vaccination period
Drowsiness (General disorders) | 17/74 | 28/95 | 34/96 | 0/0 | 33/96 — During the 4-day (Days 0-3) period following booster vaccination with Synflorix vaccine
Fever (General disorders) | 38 | 36 | 41/98 | 28/98 | 28/98 — During the 4-day (Days 0-3) post-primary vaccination period
Fever (General disorders) | 9/74 | 11/95 | 7/96 | 0/0 | 11/96 — During the 4-day (Days 0-3) period following booster vaccination with Synflorix vaccine
Irritability (General disorders) | 63 | 84 | 89/98 | 89/98 | 91/98 — During the 4-day (Days 0-3) post-primary vaccination period
Irritability (General disorders) | 25/74 | 35/95 | 31/96 | 0/0 | 43/96 — During the 4-day (Days 0-3) period following booster vaccination with Synflorix vaccine
Loss of appetite (General disorders) | 36 | 53 | 56/98 | 57/98 | 62/98 — During the 4-day (Days 0-3) post-primary vaccination period
Loss of appetite (General disorders) | 17/74 | 23/95 | 29/96 | 0/0 | 37/96 — During the 4-day (Days 0-3) period following booster vaccination with Synflorix vaccine
Pain (General disorders) | 73 | 93 | 92/98 | 95/98 | 97/98 — During the 4-day (Days 0-3) post-primary vaccination period
Pain (General disorders) | 40/74 | 58/95 | 62/96 | 0/0 | 60/96 — During the 4-day (Days 0-3) period following booster vaccination with Synflorix vaccine
Redness (General disorders) | 62 | 80 | 83/98 | 83/98 | 84/98 — During the 4-day (Days 0-3) post-primary vaccination period
Redness (General disorders) | 25/74 | 31/95 | 39/96 | 0/0 | 45/96 — During the 4-day (Days 0-3) period following booster vaccination with Synflorix vaccine
Swelling (General disorders) | 67 | 83 | 84/98 | 91/98 | 84/98 — During the 4-day (Days 0-3) post-primary vaccination period
Swelling (General disorders) | 28/74 | 39/95 | 38/96 | 0/0 | 53/96 — During the 4-day (Days 0-3) period following booster vaccination with Synflorix vaccine
Vomiting (General disorders) | 17 | 19 | 15/98 | 18/98 | 23/98 — During the 4-day (Days 0-3) post-primary vaccination period
Upper respiratory tract infection (Infections and infestations) | 4 | 13 | 13 | 11 | 12 — Within the 31-day (Days 0-30) post-primary vaccination period
Upper respiratory tract infection (Infections and infestations) | 2/76 | 5/96 | 6/98 | 0/0 | 5/98 — Within the 31-day (Days 0-30) post Synflorix booster vaccination period
Decreased appetite (Metabolism and nutrition disorders) | 4/76 | 6/96 | 4/98 | 0/0 | 4/98 — Within the 31-day (Days 0-30) post Synflorix booster vaccination period
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 73 | 67 | 58 | 66 — Within the 31-day (Days 0-30) post-primary vaccination period
Cough (Respiratory, thoracic and mediastinal disorders) | 17/76 | 23/96 | 24/98 | 0/0 | 13/98 — Within the 31-day (Days 0-30) post Synflorix booster vaccination period
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 29 | 40 | 50 | 49 | 51 — Within the 31-day (Days 0-30) post-primary vaccination period
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 7/76 | 4/96 | 6/98 | 0/0 | 6/98 — Within the 31-day (Days 0-30) post Synflorix booster vaccination period
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1/76 | 5/96 | 7/98 | 0/0 | 5/98 — Within the 31-day (Days 0-30) post Synflorix booster vaccination period
Eczema (Skin and subcutaneous tissue disorders) | 9 | 12 | 11 | 12 | 14 — Within the 31-day (Days 0-30) post-primary vaccination period
Rash (Skin and subcutaneous tissue disorders) | 26 | 25 | 16 | 28 | 21 — Within the 31-day (Days 0-30) post-primary vaccination period
Rash (Skin and subcutaneous tissue disorders) | 4/76 | 4/96 | 3/98 | 0/0 | 5/98 — Within the 31-day (Days 0-30) post Synflorix booster vaccination period
Pyrexia (General disorders) | 5 | 8 | 5 | 9 | 9 — Within the 31-day (Days 0-30) post-primary vaccination period
Bronchiolitis (Infections and infestations) | 1 | 6 | 3 | 8 | 2 — Within the 31-day (Days 0-30) post-primary vaccination period
Bronchopneumonia (Infections and infestations) | 5 | 3 | 3 | 0 | 2 — Within the 31-day (Days 0-30) post-primary vaccination period
Oral candidiasis (Infections and infestations) | 9 | 4 | 6 | 3 | 3 — Within the 31-day (Days 0-30) post-primary vaccination period
Decreased appetite (Metabolism and nutrition disorders) | 6 | 9 | 1 | 3 | 3 — Within the 31-day (Days 0-30) post-primary vaccination period
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 9 | 10 | 9 | 10 — Within the 31-day (Days 0-30) post-primary vaccination period
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 9 | 11 | 6 | 9 — Within the 31-day (Days 0-30) post-primary vaccination period
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 12 | 8 | 11 | 8 | 4 — Within the 31-day (Days 0-30) post-primary vaccination period
Eye discharge (Eye disorders) | 4 | 6 | 6 | 4 | 3 — Within the 31-day (Days 0-30) post-primary vaccination period
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 4 | 3 | 9 — Within the 31-day (Days 0-30) post-primary vaccination period
Constipation (Gastrointestinal disorders) | 0 | 3 | 3 | 5 | 6 — Within the 31-day (Days 0-30) post-primary vaccination period

LIMITATIONS AND CAVEATS:
The study aimed to enrol 100 HIV+/+ subjects but succeeded to enrol 83 mainly due to decrease of vertical HIV transmission in South Africa. Some subjects, HIV+ at screening, tested negative at subsequent HIV testing, were reallocated in HIV+/-Group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.